CLINICAL TRIAL: NCT06973876
Title: Examining the Effectiveness of Asynchronous Versus Synchronous Yoga for Veterans With Chronic Pain
Acronym: STRETCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: VHA Office of Rural Health (Unknown)
Responsible Party: Principal Investigator, Belle Zaccari, Co-Principal Investigator, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 6392 / 24-75
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Yoga
Keywords: chronic pain; yoga; synchronous telehealth; asynchronous telehealth; rural; Veterans; teleyoga
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: The research team will enroll 100 Veterans diagnosed with chronic pain to be randomized 1:1 using permuted block randomization with blocks of varying length to either synchronous teleyoga at VAPORHCS or asynchronous teleyoga via Ompractice. Virtual groups will be composed of 8-10 participants, which will require 5-7 cohorts of each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Teleyoga (Placebo Comparator): Participants randomized to receive synchronous teleyoga will be provided information so that they can attend VA Portland Health Care System (VAPORHCS) virtual yoga offerings. They will be encouraged to attend one class per week during the 12 weeks between randomization and follow-up assessment. Attendance will be tracked via a signed note in the medical record. Each session will last approximately 30-60 minutes.
  Interventions: Behavioral: Pain-Sensitive Teleyoga Primer; Behavioral: Synchronous Teleyoga
- Asynchronous Teleyoga (Active Comparator): Participants randomized to receive asynchronous teleyoga will be provided information so that they can access to the digital library of yoga videos on Ompractice, an existing partner with VA Medical Centers. Ompractice contains a suite of yoga video content, and participants will be encouraged to complete one class per week during the 12 weeks between randomization and follow-up assessment.
  Interventions: Behavioral: Pain-Sensitive Teleyoga Primer; Behavioral: Asynchronous Teleyoga

INTERVENTIONS:
Behavioral: Pain-Sensitive Teleyoga Primer — The 5-session Pain-Sensitive Teleyoga Primer will be delivered synchronously to participants who will practice from their home. The purpose of the 5-session primer is two-fold: (1) it allows trained yoga instructors to determine physical abilities and limitations of patient participants so that pose modifications may be taught and (2) it provides education to participants on pain neuroscience, breathwork, relaxation, mindfulness, and interoception so that they may apply this knowledge to maximize the benefits of whichever yoga condition they are randomized to. Each session will last approximately 75 minutes. Participants will be provided with a supplementary handout to reinforce content from the sessions.
Behavioral: Synchronous Teleyoga — Participants randomized to receive synchronous teleyoga will be provided information so that they can attend VAPORHCS virtual yoga offerings. They will be encouraged to attend one class per week during the 12 weeks between randomization and follow-up assessment. Attendance will be tracked via a signed note in the medical record. Each session will last approximately 30-60 minutes.
  Arms: Synchronous Teleyoga
Behavioral: Asynchronous Teleyoga — Participants randomized to receive asynchronous teleyoga will be provided information so that they can access to the digital library of yoga videos on Ompractice, an existing partner with VA Medical Centers. Ompractice contains a suite of yoga video content, and participants will be encouraged to complete one class per week during the 12 weeks between randomization and follow-up assessment. Attendance will be tracked by Ompractice and shared with VAPORHCS.
  Arms: Asynchronous Teleyoga

SUMMARY:
The goal of this clinical trial is to see if pre-recorded yoga videos are as helpful for chronic pain as online yoga sessions taught in real time. The main questions it aims to answer are:

Are pre-recorded yoga videos an acceptable and practical tool and could they be used more broadly?

Are pre-recorded yoga videos no worse than online yoga sessions taught in real time for managing chronic pain?

Researchers will compare changes in chronic pain, mental health, and quality of life outcomes for participants who attend pre-recorded yoga videos versus online yoga sessions taught in real time.

Over the course of 4 months, participants will:

Attend a 5-session virtual yoga course. Continue virtual yoga practice for 12-weeks on their own or in a VA online class. Complete 3 online assessments and a brief exit interview.

DETAILED DESCRIPTION:
The overarching goals of the proposed research are to pilot test feasibility and acceptability of a 5-session yoga primer to the mindful practice of pain-sensitive teleyoga and its impact on subsequent teleyoga practice delivered either synchronously or asynchronously. The research will also test the preliminary effectiveness of teleyoga practice on outcomes related to chronic pain, mental health, and quality of life.

* Aim 1: Assess acceptability and feasibility of trial methodology to inform future larger-scale trials.
* Aim 2: Use intent-to-treat analysis and random effect regression models to compare changes in pain interference, pain severity, physical function, quality of life, depression, and anxiety between participants who attend synchronous vs. asynchronous teleyoga.

The primary purpose of a pilot study is to assess feasibility of methods to inform future larger studies. However, inferential analyses may be appropriate to help ascertain estimates of variability for the primary and secondary outcomes that can be used to power larger trials. To that end, the investigators will use intent-to-treat procedures and random effect regression models to compare changes in the outcome variables between patients who receive asynchronous vs. synchronous teleyoga.

Hypothesis: The investigators predict that asynchronous teleyoga will be non-inferior to synchronous teleyoga in reducing the primary outcome of pain interference, as well as across secondary outcomes

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veteran enrolled at VAPORHCS and has established care with a VA medical or mental health provider.
* Diagnosed with musculoskeletal pain, confirmed by electronic health record review and phone screening.
* Has an average pain severity of at least 4 in the past 3 months, assessed by items 1-5 of the Brief Pain Inventory, Short Form.
* Aged 18 or over.
* Capable of using video teleconferencing to complete enrollment, assessment, and video interventions.
* Meets physical readiness, assessed by the Physical Activity Readiness Questionnaire (PAR-Q) and approved for yoga participation by their primary care team or physical therapy team.
* Able to sit and stand from the floor without assistance
* Able to ambulate community distances without an assistive device
* Intact sensation in lower extremities below the knees

Exclusion Criteria:

* Unable to read and write in English.
* Unable to freely give informed consent.
* Recent (past 3 months) psychotic symptoms consistent with a diagnosis of schizophrenia, schizoaffective disorder, delusional disorder, or other psychotic disorder and unrelated to PTSD. Assessed by medical record review and provider team.
* Practicing yoga regularly defined as weekly or biweekly practice of 60 or more minutes for 6 months or more.
* Recent (past 3 months) history of suicidal gesture related to physical pain or active suicidal ideation (plan, intent, means).
* Concurrently enrolled in another research protocol involving a pain focused intervention.
* Upcoming surgery that would impact yoga practice.
* Active alcohol/other substance abuse or dependence (unless actively engaged in treatment). Assessed via the The Tobacco, Alcohol, prescription medication and other Substance use Tool (TAPS). A cutoff of 2 will be used to rule out.
* Joint replacement within the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory Short Form (BPI-SF) | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  The Brief Pain Inventory Short Form (BPI-SF) is a widely used 9-item tool for assessing pain severity and pain interference. The primary outcome will be the Pain Interference Subscale of the BPI-SF. Scores are reported on a range of 0 - 10, with higher scores indicating more impairment due to pain.

SECONDARY OUTCOMES:
Brief Pain Inventory Short Form - Pain Severity Subscale (BPI-SF | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  Pain Severity Subscale (BPI-SF) is a widely used 9-item tool for assessing pain severity and pain interference. Scores are on a range of 0 - 10, with higher scores indicating more severe pain.
PROMIS Physical Function 4-Item Short Form Instrument | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  Physical Functioning will be assessed with the 4-item PROMIS Physical Functioning scale. The physical function form asks the participant to rate a series of physical function related questions on 5-point Likert scale, with one representing a better outcome.
Veterans RAND 12-Item Health Survey (VR-12) | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  The Veterans RAND 12-Item Health Survey (VR-12) is a 12-item instrument used to measure health related quality of life in Veterans. VR-12 scores are summarized into two scores, a Physical Health component score and a Mental Health component score. Each component score is on a range of 0 - 100, with higher scores indicating more impairment in physical or mental health, respectively.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item scale that can be used to screen, diagnose, monitor, and measure the severity of depression. The PHQ-9 scoring system ranges from 0 to 27, with higher scores indicating more severe depression
Generalized Anxiety Disorder 7-Item Scale | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  Generalized Anxiety Disorder 7-Item Scale is designed for screening and measuring the severity of generalized anxiety symptoms. Scores on the GAD-7 range from 0 - 21, with higher scores indicating more severe symptoms of anxiety.
Five-facet Mindfulness Questionnaire | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  The five-facet Mindfulness Questionnaire is a 15-item scale that measures the effectiveness of mindfulness strategies. Five subscales of mindfulness measure observing, describing, acting with awareness, non-judgment and non-reactivity. Average scores are calculated by summing the responses and dividing by the number of items, and indicate the average level of agreement with each subscale. The items use a 5-point Likert scale. Higher scores are indicative of someone who is more mindful in their everyday life.
Multidimensional Assessment of Interoceptive Awareness, Version 2 (Brief MAIA-2) | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  The Multidimensional Assessment of Interoceptive Awareness, Version 2 (Brief MAIA-2) is a 24-item scale measuring interoceptive sensibility, defined as the self-perceived tendency to focus on internal stimuli. Participants rate each item on a 6-point Likert scale, with higher scores indicating higher interoception. This measure has been shown to be reliable, including for those with a long-term health condition
PTSD Checklist for DMS-5 (PCL-5) | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  The PTSD Checklist for DMS-5 (PCL-5) is a 20-item self-report questionnaire that assesses the severity of symptoms associated with exposure to trauma. Participants rate 20 items in the past month on a 5- point Likert scale. Total scores range from 0 (best outcome) to 80 (worst outcome).
Well-Being Signs | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  Well-Being Signs is a three-question screening tool used to assess how Veterans are doing in their daily lives. Each question uses a 10-point Likert scale. An average score is calculated based on the ratings for each of the questions with higher scores indicating better well-being.
Pain Catastrophizing Scale | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  Pain Catastrophizing Scale measures catastrophizing related to chronic pain and is used extensively in clinical practice and in research. The pain catastrophizing scale consists of 13 items These are divided into 3 domains: rumination, magnification and helplessness. The subject is asked to indicate how how well each sentence applies for them on a 4-point Likert scale. The total score on the questionnaire can lie between 0 - 52 where a higher score indicates higher levels of pain catastrophizing thoughts.
Teleyoga Attendance and Engagement (EHR & Digital Well-Being Data Collection) | Baseline, Post 5-session Yoga Primer (Week 5/6), Week 18
  Attendance and engagement during the Yoga Primer and each intervention arm will be collected. Virtual yoga completed as part of the 5-session primer and in the Synchronous Teleyoga arm will be documented via a note attached and have a visit assigned as well to chart on in the medical record. Attendance and engagement in the Asynchronous Teleyoga arm will be documented and tracked through Ompractice through participant internet protocol address, which participants consent to sharing when they sign up and read the terms of use.

OTHER OUTCOMES:
Semi-structured interview | Week 18
  Semi-structured interviews will be conducted following the final online data collection. Interviews will be used to collect additional feedback about the intervention and data collection experience. Rapid Qualitative Analysis will be used to analyze semi-structured interview data.

CONTACTS AND LOCATIONS:
Locations (1):
- Portland VA Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No